CLINICAL TRIAL: NCT04232371
Title: Randomized Clinical Trial for Treatment of Atrioventricular Nodal Reentry Tachycardia (AVNRT): Low Voltage and Wave Front Collision Mapping vs. Anatomic/Electrogram Approach to Slow AV Nodal Pathway Ablation
Brief Title: Treatment Study of AV Node Reentry Tachycardia
Acronym: AVNRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeffrey Moak (Other)
Collaborators: University of Iowa (Other); University of Wisconsin, Madison (Other); University of Louisville (Other); Memorial Health System (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Moak, Director, Electrophysiology and Pacing, Principal Investigator, Clinical Professor, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011178
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Supraventricular Tachycardia
Keywords: New Ablation Technique; Standard Ablation Technique
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Intervention Model Description: Patients will be randomized within each participating center, not by center, into study groups:
  1. New Ablation Technique - will undergo ablation using voltage mapping and triangle of Koch propagation wave collision mapping. Ablation will be performed at or slightly above the site of wave front collision.
  2. Standard Ablation Technique - ablation performed using the traditional anatomical / electrogram guided ablation approach.
  Randomization will occur through a module in Redcap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- New Ablation Technique (Active Comparator): Will undergo ablation using voltage mapping and triangle of Koch propagation wave collision mapping. Ablation will be performed at or slightly above the site of wave front collision.
  Interventions: Procedure: New Ablation Technique
- Standard Ablation Technique (Active Comparator): Ablation performed using the traditional anatomical / electrogram guided ablation approach.
  Interventions: Procedure: Standard Ablation Technique

INTERVENTIONS:
Procedure: New Ablation Technique — Patient will undergo ablation using voltage mapping and triangle of Koch propagation wave collision mapping. Ablation will be performed at or slightly above the site of wave front collision.
  Arms: New Ablation Technique
Procedure: Standard Ablation Technique — Ablation performed using the traditional anatomical / electrogram guided ablation approach.
  Arms: Standard Ablation Technique

SUMMARY:
Compare the effectiveness and safety of two techniques for modification of slow AV nodal pathway conduction underlying AVNRT: 1) New Ablation Technique, low voltage and wave front collision mapping vs. 2) the Standard Ablation Technique, an anatomical/electrogram approach.

DETAILED DESCRIPTION:
Supraventricular tachycardia (SVT) is an arrhythmia condition that affects 1 in 250 to 1/1000 children. While there are many different mechanisms for SVT, having an additional electrical pathway in the heart is the most common underlying reason. The extra electrical pathway may be in the form of an accessory AV pathway that bridges the atrium and ventricle or a slowing conducting pathway in the AV nodal region. SVT may cause significant disability from the sudden unexpected rapid increase in heart rate. Symptoms associated with SVT may include dizziness, syncope, shortness of breath, chest pain and exercise intolerance. Prolonged episodes that do not self terminate may require the patient to be evaluated in an emergency room. If left untreated, SVT may result in congestive heart failure and the potential for sudden cardiac arrest.

Catheter based ablation involves the localized application of energy to the site responsible for the SVT, effecting a permanent cure. Ablation has become the primary mode for treating patients with SVT. Ablation is achieved by the focal and limited application of energy (either heating the tissue to temperatures beyond viability, radiofrequency energy (RF)) or cooling the tissue (cryoablation)) to functionally destroy the underlying myocardial tissue. Both energy sources are very effective in achieving this end point, and the elimination of arrhythmias.

SVT involving the AV node, known as AV node reentry tachycardia (AVNRT), is one of the most common forms of this arrhythmia. While a conceptual construct for understanding AV node reentry tachycardia has evolved over the years, the subtleties of the exact pathophysiologic mechanism leading to its occurrence is undefined. Most of the medical literature endorses the concept of two (dual) inputs into the compact AV node. Circus movement or reentry incorporating the fast and slow pathways (two AV nodal pathways) is thought to facilitate this form of SVT. Current ablation practice is centered on modification of the slow AV nodal pathway conduction, leaving the fast AV nodal pathway intact so as to allow for a normal conduction interval between the atrium and ventricule, the PR interval.

Approaches for ablation of the slow AV nodal pathway differ among pediatric centers. The two most used techniques for ablation of the slow AV nodal pathway to prevent AV nodal reentry tachycardia involve: 1) an anatomical/electrogram approach based on physical position of the ablation catheter and the electrogram morpholog (Standard Technique), and 2) mapping of electrogram voltage in the triangle of Koch to define an area of low voltage with assessment of the site for wave front collision of electrical activity traveling over the fast and slow AV nodal pathways (New Technique).

ELIGIBILITY:
Inclusion Criteria:

1. Weight >15 kg
2. Age < 21 years old
3. Simple CHD acceptable to enroll (Table 1):

Table 1. Diagnoses in Adult Patients with Simple Congenital Heart Disease

* Isolated congenital aortic valve disease
* Isolated congenital mitral valve disease (eg, except parachute valve, cleft leaflet)
* Small atrial septal defect
* Isolated small ventricular septal defect (no associated lesions)
* Mild pulmonary stenosis
* Small patent ductus arteriosus
* Repaired conditions
* Previously ligated or occluded ductus arteriosus
* Repaired secundum or sinus venosus atrial septal defect without residua
* Repaired ventricular septal defect without residua

Exclusion Criteria:

1. Additional mechanism(s) for SVT in addition to AV nodal reentry tachycardia.
2. Moderate or Complex Congenital Heart Disease, see tables 2 and 3.

Table 2. Diagnoses in Adult Patients with Congenital Heart Disease of Moderate Complexity

* Aorto-left ventricular fistulas
* Anomalous pulmonary venous drainage, partial or total
* Atrioventricular septal defects (partial or complete)
* Coarctation of the aorta
* Ebstein's anomaly
* Infundibular right ventricular outflow obstruction of significance
* Ostium primum atrial septal defect
* Patent ductus arteriosus (not closed)
* Pulmonary valve regurgitation (moderate to severe)
* Pulmonary valve stenosis (moderate to severe)
* Sinus of Valsalva fistula/aneurysm
* Sinus venosus atrial septal defect
* Subvalvular AS or SupraAS (except HOCM)
* Tetralogy of Fallot
* Ventricular septal defect with:
* Absent valve or valves
* Aortic regurgitation
* Coarctation of the aorta
* Mitral disease
* Right ventricular outflow tract obstruction
* Straddling tricuspid/mitral valve
* Subaortic stenosis

Table 3. Types of Adult Congenital Heart Disease - Severe Complexity

* Conduits, valved or nonvalved
* Cyanotic congenital heart (all forms)
* Double-outlet ventricle
* Eisenmenger syndrome
* Fontan procedure
* Mitral atresia
* Single ventricle (also called double inlet or outlet, common, or primitive)
* Pulmonary atresia (all forms)
* Pulmonary vascular obstructive disease
* Transposition of the great arteries
* Tricuspid atresia
* Truncus arteriosus/hemitruncus
* Other abnormalities of atrioventricular or ventriculoarterial connection not included above (ie, crisscross heart, isomerism, heterotaxy syndromes, ventricular inversion)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Primary end point - Number of lesions needed to achieve modification of slow AV nodal pathway | During procedure- start to finish
  Number of ablation lesion needed to achieve modification of slow AV nodal pathway conduction underlying AVNRT as defined by one of the following:
  1. Absent SVT induction
  2. Loss of slow pathway function as defined by no jumps (discontinuity in AV conduction curve) or unable to sustain PR > RR during rapid atrial pacing
  3. Persistence of dual pathway physiology with no echo beat
  4. Persistence of dual pathway physiology with single echo beat

SECONDARY OUTCOMES:
Secondary End points - Time from start to end of ablation lesion application(s), and total length of procedure. | During procedure- start to finish
  1. Time from start to end of ablation lesion application(s)
  2. Procedure time (sheath in to time of final sheath removal)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moak, Principal Investigator — Children's National Research Institute
Locations (5):
- United States (5):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Memorial Health System, Hollywood, Florida
  - Univeristy of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Philip Saul J, Kanter RJ; WRITING COMMITTEE; Abrams D, Asirvatham S, Bar-Cohen Y, Blaufox AD, Cannon B, Clark J, Dick M, Freter A, Kertesz NJ, Kirsh JA, Kugler J, LaPage M, McGowan FX, Miyake CY, Nathan A, Papagiannis J, Paul T, Pflaumer A, Skanes AC, Stevenson WG, Von Bergen N, Zimmerman F. PACES/HRS expert consensus statement on the use of catheter ablation in children and patients with congenital heart disease: Developed in partnership with the Pediatric and Congenital Electrophysiology Society (PACES) and the Heart Rhythm Society (HRS). Endorsed by the governing bodies of PACES, HRS, the American Academy of Pediatrics (AAP), the American Heart Association (AHA), and the Association for European Pediatric and Congenital Cardiology (AEPC). Heart Rhythm. 2016 Jun;13(6):e251-89. doi: 10.1016/j.hrthm.2016.02.009. Epub 2016 Feb 17. No abstract available. PMID 26899545
- [Background] Papagiannis J, Beissel DJ, Krause U, Cabrera M, Telishevska M, Seslar S, Johnsrude C, Anderson C, Tisma-Dupanovic S, Connelly D, Avramidis D, Carter C, Kornyei L, Law I, Von Bergen N, Janusek J, Silva J, Rosenthal E, Willcox M, Kubus P, Hessling G, Paul T; Pediatric and Congenital Electrophysiology Society. Atrioventricular Nodal Reentrant Tachycardia in Patients With Congenital Heart Disease: Outcome After Catheter Ablation. Circ Arrhythm Electrophysiol. 2017 Jul;10(7):e004869. doi: 10.1161/CIRCEP.116.004869. Epub 2017 Jul 7. PMID 28687669
- [Background] Markowitz SM, Lerman BB. A contemporary view of atrioventricular nodal physiology. J Interv Card Electrophysiol. 2018 Aug;52(3):271-279. doi: 10.1007/s10840-018-0392-5. Epub 2018 Jun 16. PMID 29909540
- [Background] Lee PC, Chen SA, Hwang B. Atrioventricular node anatomy and physiology: implications for ablation of atrioventricular nodal reentrant tachycardia. Curr Opin Cardiol. 2009 Mar;24(2):105-12. doi: 10.1097/HCO.0b013e328323d83f. PMID 19225293
- [Background] Malloy L, Law IH, Von Bergen NH. Voltage mapping for slow-pathway visualization and ablation of atrioventricular nodal reentry tachycardia in pediatric and young adult patients. Pediatr Cardiol. 2014 Jan;35(1):103-7. doi: 10.1007/s00246-013-0748-7. Epub 2013 Jul 20. PMID 23872907
- [Background] Van Aartsen A, Law IH, Maldonado JR, Von Bergen NH. Propagation Mapping Wave Collision Correlates to the Site of Successful Ablation During Voltage Mapping in Atrioventricular Nodal Reentry Tachycardia. J Innov Card Rhythm Manag. 2017 Sep 15;8(9):2836-2842. doi: 10.19102/icrm.2017.080905. eCollection 2017 Sep. PMID 32494469
- [Background] Collins KK, Dubin AM, Chiesa NA, Avasarala K, Van Hare GF. Cryoablation versus radiofrequency ablation for treatment of pediatric atrioventricular nodal reentrant tachycardia: initial experience with 4-mm cryocatheter. Heart Rhythm. 2006 May;3(5):564-70. doi: 10.1016/j.hrthm.2006.01.026. Epub 2006 Feb 28. PMID 16648062
- [Background] Kammeraad J, Udink ten Cate F, Simmers T, Emmel M, Wittkampf FH, Sreeram N. Radiofrequency catheter ablation of atrioventricular nodal reentrant tachycardia in children aided by the LocaLisa mapping system. Europace. 2004 May;6(3):209-14. doi: 10.1016/j.eupc.2004.02.004. PMID 15121072
- [Background] Kriebel T, Bertram H, Windhagen-Mahnert B, Bokenkamp R, Kaulitz R, Rohloff A, Peuster M, Hausdorf G, Paul T. [Atrioventricular nodal reentry tachycardia in children: curative treatment by high frequency catheter ablation]. Z Kardiol. 2000 Jun;89(6):538-45. doi: 10.1007/s003920070226. German. PMID 10929439
- [Background] Rhodes LA, Wieand TS, Vetter VL. Low temperature and low energy radiofrequency modification of atrioventricular nodal slow pathways in pediatric patients. Pacing Clin Electrophysiol. 1999 Jul;22(7):1071-8. doi: 10.1111/j.1540-8159.1999.tb00572.x. PMID 10456636
- [Background] Teixeira OH, Balaji S, Case CL, Gillette PC. Radiofrequency catheter ablation of atrioventricular nodal reentrant tachycardia in children. Pacing Clin Electrophysiol. 1994 Oct;17(10):1621-6. doi: 10.1111/j.1540-8159.1994.tb02355.x. PMID 7800563
- [Background] Papagiannis J, Papadopoulou K, Rammos S, Katritsis D. Cryoablation versus radiofrequency ablation for atrioventricular nodal reentrant tachycardia in children: long-term results. Hellenic J Cardiol. 2010 Mar-Apr;51(2):122-6. PMID 20378513
- [Background] PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.
- [Background] Chow, S.C.; Shao, J.; Wang, H. 2003. Sample Size Calculations in Clinical Research. Marcel Dekker. New York.